CLINICAL TRIAL: NCT05623501
Title: Phase I, Dose-Escalation Study of Dihydromyricetin (DHM) to Treat Alcohol-Associated Liver Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Brian P. Lee, Assistant Professor of Medicine, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-00428
Record Dates: First submitted 2022-11-11; First posted 2022-11-21 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Alcohol-Related Disorders
MeSH Terms: conditions — Alcohol-Related Disorders | interventions — dihydromyricetin

STUDY DESIGN:
Intervention Model Description: This is a single-center dose-escalation study. A total of 12 participants are planned and will be divided into 4 cohorts with 3 participants per cohort. Cohort 1 will consist of three healthy volunteers who will receive DHM in two doses of 300 mg as liquid suspension. Cohort 2 will consist of three healthy volunteers who will receive DHM in two doses of 900 mg as liquid suspension. Cohort 3 will consist of three healthy volunteers who will receive DHM in two 50mL PO solution doses of 300 mg plus 140mg L-lysine. Cohort 4 will consist of three healthy volunteers who will receive DHM in two 50mL PO solution doses of 900 mg plus 420mg L-lysine. Each participant will be administered the study drug during a 24-hour period, requiring two consecutive days of visits to research clinic. Evaluations will be taken at uniform intervals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): DHM 300mg x1 dose
  Interventions: Drug: Dihydromyricetin
- Cohort 2 (Experimental): DHM 900mg x1 dose
  Interventions: Drug: Dihydromyricetin
- Cohort 3 (Experimental): DHM 300mg x1 dose + Lysine 140mg x1 dose
  Interventions: Drug: Dihydromyricetin
- Cohort 4 (Experimental): DHM 900mg x1 dose + Lysine 420mg x1 dose
  Interventions: Drug: Dihydromyricetin

INTERVENTIONS:
Drug: Dihydromyricetin — Dose-escalation and lysine preparation

SUMMARY:
The current proposal is designed as a first-in-human Phase 1 open-label, dose-escalation study to assess the safety, pharmacokinetics, and the maximum tolerated dose of DHM among healthy volunteers using a purified form of DHM from a local cGMP compliant source (Master Herbs, Inc).

DETAILED DESCRIPTION:
Dihydromyricetin (DHM), a bioactive flavonoid from an edible plant (ampelopsis grossedentata), is reported to have multiple protective effects against chemical-induced liver injuries. For example, the antioxidant activity and cellular metabolic protective effects of DHM may act via the AMP kinase (AMPK) and nicotinamide adenine dinucleotide (NAD+)-dependent Sirtuin (Sirt)-1 energy regulating pathway. Furthermore, there is accumulating evidence supporting the use of DHM for the treatment of alcohol use disorder and the possible reduction/prevention of alcohol-associated liver disease in animal models. DHM may represent a novel approach to counteract alcohol-induced liver damage and promote alcohol metabolism via changes in hepatocellular bioenergetics and mitochondrial biogenesis driven by the AMPK/Sirt-1/PGC-1α axis.

These preclinical data suggest the potential of DHM as a novel therapeutic agent in alcohol-related diseases. However, further study in humans is warranted. While DHM has been used for herbal tea in traditional Chinese medicine for hundreds of years, and there has been a small clinical trial using DHM in China among individuals with non-alcoholic fatty liver disease, there have been no controlled human studies published that have assessed the safety, pharmacokinetics, or optimal dosing of DHM in humans.

DHM is marketed as a dietary supplement in the United States and is not regulated by the Food and Drug Administration (FDA) as a drug. Because the FDA has little control over the quality of herbal products such as DHM, it is necessary to quantitatively estimate the potentially active ingredients and the pharmacokinetic (PK) profile with oral administration.

The current proposal is designed as a first-in-human Phase 1 open-label, dose-escalation study to assess the safety, pharmacokinetics, and the maximum tolerated dose of DHM among healthy volunteers using a purified form of DHM from a local cGMP compliant source (Master Herbs, Inc).

ELIGIBILITY:
Inclusion Criteria:

* No prior medical history of alcohol use disorder or alcohol-associated liver disease
* Between 18-60 years old

Exclusion Criteria:

* Weight below 50kg.
* Advanced liver disease
* Other acute liver diseases
* HIV co-infection
* History of pancreatic or biliary disease
* Acute illness that would interfere with drug absorption
* Pregnancy
* Participants who are currently taking drugs with CYP3A4 effects
* FIB-4 Index > 1.30
* History of Alcohol Use Disorder (AUD) determined by score > 8 on AUDIT questionnaire

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic of DHM | -0.5 (pre-dose), 0 (1st dose), 0.5, 1, 2, 4, 6, 8 (2nd dose), 10, and 24 hours post-dose.
  serum DHM metabolites will be performed using MRM mass
Adverse Events | 24 hours post-dose
  The National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 will be used to assess and grade AE severity

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lee, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Undecided